CLINICAL TRIAL: NCT02012127
Title: Description of Sign-and-symptom Associations at Acromegaly Diagnosis.
Acronym: ACRO-POLIS
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-54-52030-266
Record Dates: First submitted 2013-11-28; First posted 2013-12-16 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Acromegalic patients

SUMMARY:
The purpose of this study is to describe most characteristic association of signs and symptoms present at the time of acromegaly diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (greater than or equal to 18 years old)
* Patient with acromegaly, diagnosed for less than 5 years

Exclusion Criteria:

* Patient who have objected to the collection of his/her data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acromegalic patients
Sampling Method: Probability Sample
Enrollment: 648 (Actual)
Dates: Start 2013-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Description of the most characteristic sign-and-symptom associations of acromegaly, collected by a patient questionnaire. | At the time of patient diagnosis, up to 3 months

SECONDARY OUTCOMES:
Description of demographic and clinical characteristics of patients with acromegaly, collected by a patient questionnaire. | At the time of patient diagnosis, up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (25):
- France (25):
  - Hôpital Sud, Amiens
  - CHU Besançon Hôpital Jean Minjoz, Besançon
  - Hôpital la Cavale Blanche, Brest
  - Chu Cote de Nacre, Caen
  - Hôpital Henri Mondor, Créteil
  - Chu de Grenoble Hôpital Albert Michallon, Grenoble
  - Hôpital Claude Huriez, Lille
  - Hôpital le Cluzeau, Limoges
  - Hôpital Neuro-cardiologique, Lyon
  - Hôpital de la Timone, Marseille
  - Hôpital Lepeyronie, Montpellier
  - Hôpitaux de Brabois, Nancy
  - CHR Orléans - Hôpital la Source, Orléans
  - CH de Bicetre, Paris
  - CH Pitie Salpetreire, Paris
  - Hôpital Lariboisiere, Paris
  - Hôpital Haut Leveque, Pessac
  - CHU Reims - Hôpital Robert Debre, Reims
  - Hôpital Sud Anne de Bretagne, Rennes
  - CHU Rouen - Hôpital de Bois Guillaume, Rouen
  - Hôptital Nord, Saint-Etienne
  - Hôpital Civil, Strasbourg
  - Hôpital de Hautepierre, Strasbourg
  - Hôpital Larrey, Toulouse
  - CHU Bretonneau, Tours

REFERENCES:
- [Derived] Caron P, Brue T, Raverot G, Tabarin A, Cailleux A, Delemer B, Renoult PP, Houchard A, Elaraki F, Chanson P. Signs and symptoms of acromegaly at diagnosis: the physician's and the patient's perspectives in the ACRO-POLIS study. Endocrine. 2019 Jan;63(1):120-129. doi: 10.1007/s12020-018-1764-4. Epub 2018 Sep 29. PMID 30269264